CLINICAL TRIAL: NCT03796013
Title: A Randomized, Open-Label, Two-Treatment, Two-Period, Two-Way Crossover Study to Investigate the Bioequivalence of Entrectinib Polymorph Forms A and C Under Fasted Conditions in Healthy Subjects
Brief Title: A Study to Investigate the Bioequivalence of Two Different Forms of Entrectinib (Forms A and C) Under Fasted Conditions in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GP41049
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Results first posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Form A to Form C Crossover (Experimental): Participants first randomized to this arm will receive a single oral dose of entrectinib form A (reference form) under fasted conditions on Day 1 of each Period. This dose will be followed by a minimum 14-day washout period, after which participants will receive a single oral dose of entrectinib form C (test form) under fasted conditions on Day 1 of Period 2 (Periods 1 and 2 = 6 days).
  Interventions: Drug: Entrectinib Form A; Drug: Entrectinib Form C
- Form C to Form A Crossover (Experimental): Participants first randomized to this arm will receive a single oral dose of entrectinib form C (test form) under fasted conditions on Day 1 of each Period. This dose will be followed by a minimum 14-day washout period, after which participants will receive a single oral dose of entrectinib form A (reference form) under fasted conditions on Day 1 of Period 2 (Periods 1 and 2 = 6 days).
  Interventions: Drug: Entrectinib Form A; Drug: Entrectinib Form C

INTERVENTIONS:
Drug: Entrectinib Form A — Participants will receive a single oral dose of entrectinib form A under fasted conditions.
Drug: Entrectinib Form C — Participants will receive a single oral dose of entrectinib form C under fasted conditions.

SUMMARY:
This study aims to demonstrate similarities between two different forms of entrectinib (A and C) when administered under fasted conditions in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy in the opinion of the investigator. Healthy is defined by the absence of evidence of any active disease or clinically significant medical condition based on a detailed medical history and examination
* Negative test results for Hepatitis B, Hepatitis C, and Human Immunodeficiency Virus (HIV)
* Females must not be pregnant or breastfeeding, and females of childbearing potential will agree to use highly-effective contraception. Females of childbearing potential must also agree to refrain from donating eggs during the treatment period and for 6 weeks after the final dose of study drug
* Males must agree to use contraception and to refrain from sperm donation from check-in (Day -1 of Period 1) to 90 days after the final dose of study drug

Exclusion Criteria:

* History of gastrointestinal surgery or other gastrointestinal disorder that might affect absorption of medicines from the gastrointestinal tract
* Presence of a clinically significant disease, illness, medical condition or disorder, or any other medical history determined by the investigator to be clinically significant and relevant. Ongoing chronic disorders which are not considered clinically significant are permissible providing they are stable
* Clinically significant change in health status, as judged by the investigator, or any major illness within the 4 weeks before screening, or clinically significant acute infection or febrile illness within the 14 days before screening
* Participation in any other clinical study involving an investigational medicinal product (IMP) or device within 30 days or 5 half-lives (if known), whichever is longer, before screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Covance Research Unit - Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Form A to Form C Crossover: Participants first randomized to this arm received a single oral dose of entrectinib form A (reference form) under fasted conditions on Day 1 of Period 1. This dose was followed by a minimum 14-day washout period, after which participants received a single oral dose of entrectinib form C (test form) under fasted conditions on Day 1 of Period 2 (Periods 1 and 2 = 6 days).
- Form C to Form A Crossover: Participants first randomized to this arm received a single oral dose of entrectinib form C (test form) under fasted conditions on Day 1 of Period 1. This dose was followed by a minimum 14-day washout period, after which participants received a single oral dose of entrectinib form A (reference form) under fasted conditions on Day 1 of Period 2 (Periods 1 and 2 = 6 days).
Period: Period 1
Arm/Group | Form A to Form C Crossover | Form C to Form A Crossover
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Form A to Form C Crossover | Form C to Form A Crossover
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Form A to Form C Crossover | Form C to Form A Crossover | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (8.4) | 44.4 (11.7) | 44 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 8 | 9 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 8 | 16
  Black or African American | 5 | 5 | 10
  Asian | 0 | 1 | 1
  Multiple | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve (AUC0-t) of Entrectinib and M5 Metabolite
Time Frame: At pre-defined intervals from Hour 0 through Day 5 of each study Period (Periods 1 and 2 = 6 days)
Population: The PK Population consisted of all participants who received at least 1 dose of study drug and had at least 1 evaluable postdose pharmacokinetic (PK) sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Form A Reference Formulation: Participants who received a single oral dose of entrectinib form A (reference form) under fasted conditions on Day 1 of Period 1 and Day 1 of Period 2 (Periods 1 and 2 = 6 days).
- Form C Test Formulation: Participants who received a single oral dose of entrectinib form C (test form) under fasted conditions on Day 1 of Period 1 and Day 1 of Period 2 (Periods 1 and 2 = 6 days).
Arm/Group | Form A Reference Formulation | Form C Test Formulation
Number analyzed (Participants) | 28 | 28
nmol*h/L
  Entrectinib | 18500 (37.9) | 16600 (30.7)
  M5 metabolite | 3610 (37.0) | 3070 (36.9)

2. Primary Outcome: Maximum Observed Concentration (Cmax) of Entrectinib and M5 Metabolite
Time Frame: At pre-defined intervals from Hour 0 through Day 5 of each study Period (Periods 1 and 2 = 6 days)
Population: The PK Population consisted of all participants who received at least 1 dose of study drug and had at least 1 evaluable postdose PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Form A Reference Formulation | Form C Test Formulation
Number analyzed (Participants) | 28 | 28
nmol/L
  Entrectinib | 796 (35.6) | 726 (28.9)
  M5 metabolite | 138 (47.9) | 114 (50.3)

3. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline through the end of study (up to clinical cut-off date 06 Feb 2019 [28 days])
Population: The Safety Population consisted of all participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Form A Reference Formulation | Form C Test Formulation
Number analyzed (Participants) | 28 | 28
Percentage of Participants | 7.1 | 0

ADVERSE EVENTS:
Time Frame: Baseline through the end of study (up to clinical cut-off date 06 Feb 2019 [28 days])
Description: The Safety Population consisted of all participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Arm/Group | Form A Reference Formulation | Form C Test Formulation
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 2/28 | 0/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Form A Reference Formulation (N=28) | Form C Test Formulation (N=28)
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT03796013/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/13/NCT03796013/SAP_001.pdf